CLINICAL TRIAL: NCT06136572
Title: Epidemiology of Assertiveness and Emotion Management Disorders in People With Tourette's Syndrome
Acronym: AFFIRMATICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RNI 2023 JALENQUES
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rathus Assertiveness scale (Experimental): All participants
  Interventions: Diagnostic Test: Rathus Assertiveness scale

INTERVENTIONS:
Diagnostic Test: Rathus Assertiveness scale — Questionnaire completion

SUMMARY:
The goal of this study is to evaluate the proportion of assertiveness difficulties in Tourette syndrome. Participants will complete several e-questionnaires (on assertiveness, Tourette severity, quality of life, self-esteem and comorbidities like depression, anxiety...).

ELIGIBILITY:
Inclusion Criteria:

* Tourette syndrome
* Participants aged 18 years or over

Exclusion Criteria:

* Participants under legal protection
* Inability to complete questionnaires alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Rathus assertiveness questionnaire | 5 minutes at inclusion
  The Rathus assertiveness questionnaire includes 30 items, each scores from -3 to +30. A total score inferior or equal to -9 reveals assertiveness difficulties.

SECONDARY OUTCOMES:
MOVES | less than 5 minutes at inclusion
  The MOVES is a self-questionnaire including 20 items which measures the severity of the Tourette syndrome. Several scores are defined : motor tics, vocal tics, obsession, compulsion and other phenomena. The higher the score, the greater the severity.
HADS | 3 minutes at inclusion
  The HADS is a self-questionnaire to assess depression (7 items) and anxiety (7 items).
ASRS-5 | 2 minutes at inclusion
  The Adult AD-HD Self-Report Scale (ASRS-5) is a scale to assess the presence of Attention-Deficit / Hyperactivity Disorder. We used the first 6 items of the questionnaire for the screening of ADHD. The total score ranges from 0 to 24 and a cut off of 13 shows good screening performance.
Rosenberg Self-Esteem Scale | 2-3 minutes at inclusion
  The Rosenberg Self-Esteem Scale is a self-questionnaire on self-esteem. It includes 10 items. The lower the score, the lower the self-esteem.
DERS | 5 minutes at inclusion
  The Difficulties in Emotion Regulation Scale (DERS) is a self-questionnaire including 36 items. Lower scores indicate the presence of difficulties in emotion regulation.
GTS-QoL | 5 minutes at inclusion
  The GTS-QoL is a specific Gilles de la Tourette Syndrome Quality of Life Scale. It consists of 27 items giving 6 dimensions: "Psychological", "Physical and activities of daily life", "Obsessive-compulsive", "Cognitive", "Social" and "Echo-coprophenomena", scored out of 100. The scores the highest represent a poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle JALENQUES, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No